CLINICAL TRIAL: NCT07110064
Title: Iparomlimab and Tuvonralimab Injection (QL1706) in Combination With Lenvatinib and AG Regimen as First-line Treatment for Advanced Metastatic Pancreatic Cancer:A Prospective, Single-Arm, Multicenter, Phase II Clinical Study
Brief Title: QL1706+Lenvatinib+AG Regimen as First-line Treatment for Advanced Metastatic Pancreatic Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Du Juan (Other)
Responsible Party: Sponsor-Investigator, Du Juan, Nanjing Drum Tower Hospital, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Organization: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-0462-02
Record Dates: First submitted 2025-07-31; First posted 2025-08-07 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Advance Pancreatic Cancer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- QL1706+Lenvatinib+AG Regimen (Experimental)
  Interventions: Drug: QL1706+Lenvatinib+AG Regimen

INTERVENTIONS:
Drug: QL1706+Lenvatinib+AG Regimen — Participants will receive QL1706 combination with Lenvatinib and AG regimen for 8 cycles. Subsequently, the enrolled patients will continue to receive maintenance therapy with QL1706 and Lenvatinib until disease progression (PD) is observed, intolerable adverse events occur, or the investigator deems it inappropriate for the subject to continue treatment.

SUMMARY:
The investigators plan to initiate a prospective, multicenter, phase II study, recruiting 80 patients with advanced pancreatic cancer who have not received prior treatment. This study aims to enhance the anti-tumor immune effect through the combination of QL1706+Lenvatinib+AG regimen, thereby improving the prognosis of patients with advanced metastatic pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* a. Age ≥18 years, ECOG performance status ≤2, and expected survival of ≥3 months.
* b. Patients with histologically or cytologically confirmed advanced metastatic pancreatic cancer.
* c. At least one measurable lesion according to RECIST 1.1 criteria;
* d. No prior anti-tumor treatment of any kind.
* e. Patients must meet the following hematological criteria: e1. White blood cell count (WBC) ≥3.0×10^9/L; e2. Absolute neutrophil count (ANC) ≥1.5×10^9/L; e3. Hemoglobin (HB) ≥90 g/L; e4. Platelet count (PLT) ≥75×10^9/L; e5. Total bilirubin (TBIL) ≤1.5× upper limit of normal (ULN); e6. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5×ULN; if there is liver metastasis, then ALT and AST ≤5×ULN; e7. Serum creatinine (Cr) ≤1×ULN or creatinine clearance (CCr) ≥50 ml/min;
* f. Doppler ultrasound assessment: Left ventricular ejection fraction (LVEF) ≥ lower limit of normal (50%).
* g. Patients of childbearing potential must take appropriate protective measures (contraception or other methods of fertility control) before enrollment and during the study.
* h. Willingness to participate in the study, with signed informed consent, good compliance, and cooperation with follow-up; able to adhere to the study protocol and follow-up procedures.

Exclusion Criteria:

* a. Prior receipt of systemic anti-tumor treatment, such as chemotherapy, radiotherapy, or other anti-tumor treatments.
* b. Participation in another drug clinical trial within the past 4 weeks.
* c. Subjects who, in the investigator's judgment, have the opportunity for surgery or are potentially operable (subjects who voluntarily forgo surgical treatment may be enrolled after investigator assessment and agreement).
* d. Subjects with moderate ascites requiring drainage (except for those with minimal ascites shown on imaging without symptoms).
* e. Known symptomatic central nervous system metastases and/or carcinomatous meningitis.
* f. History of other primary malignancies, except for the following: 1) Malignancies that have been in complete remission for at least 2 years prior to enrollment and do not require other treatments during the study; 2) Non-melanoma skin cancer or malignant lentigo that has been adequately treated and shows no evidence of disease recurrence; 3) Carcinoma in situ that has been adequately treated and shows no evidence of disease recurrence.
* g. Patients with autoimmune diseases or immune deficiencies who are being treated with immunosuppressive drugs.
* h. Patients with a tendency to bleed.
* i. Pregnant or breastfeeding women. Women of childbearing potential must have a negative pregnancy test within 7 days prior to enrollment.
* j. Drug abuse, or clinical, psychological, or social factors that may affect informed consent or study implementation.
* k. Subjects who may be allergic to epaltrastide (QL1706), lenvatinib, albumin-bound paclitaxel, or gemcitabine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-09-03 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Median Progression-Free Survival (mPFS) | up to 24 months

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | up to 24 months
Disease Control Rate (DCR) | up to 24 months
Median Overall Survival (mOS) | up to 24 months
Adverse Events（AEs） | up to 36 months

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing Drum Tower Hospital, Nanjing, China

IPD SHARING:
Plan to Share IPD: No